CLINICAL TRIAL: NCT02763397
Title: Deep Brain Stimulation (DBS) of the Nucleus Basalis of Meynert (NbM) in Patients With Parkinson's Disease: A Pilot Study
Brief Title: Deep Brain Stimulation (DBS) of the Nucleus Basalis of Meynert (NbM) in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Teus van Laar, Prof. Dr., University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL 57011.042.16
Record Dates: First submitted 2016-04-27; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Cognitive Deficit
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- NBM-DBS on (Experimental): DBS is programmed to stimulate the NbM
  Interventions: Device: NBM-DBS
- DBS off (Placebo Comparator): DBS is turned off, no stimulation will be exerted
  Interventions: Device: DBS

INTERVENTIONS:
Device: NBM-DBS — DBS which has already been implanted aiming initially to stimulate the GPi will be reprogrammed in order to stimulate more distal structure, the NBM.
  Arms: NBM-DBS on
Device: DBS — DBS will be switched off
  Arms: DBS off

SUMMARY:
The existing DBS setting in patients with DBS of the globus pallidus interna (GPi), which aims to treat motor symptoms by a high-frequency stimulation, will be temporarily reprogramed to stimulate the NbM at a low frequency using the distal electrodes positioned in the vicinity of the NBM.

This study aims to investigate the neuropsychological effect of low frequency stimulation of the nucleus basalis of Meynert (NBM) in advanced Parkinson's disease (PD) patients, who were previously treated with deep brain stimulation (DBS) of the globus pallidus interna (GPi).

DETAILED DESCRIPTION:
The existing DBS setting in patients with GPi DBS, which aims to treat motor symptoms by a high-frequency stimulation, will be temporarily reprogramed to stimulate the NBM at a low frequency using the distal electrodes positioned in the vicinity of the NBM.This study consists of a three-day screening study of the NbM stimulation followed by a two-week, randomized, single-blind, crossover trial. Between the screening study and the crossover trial, one week of washout period will be applied to eliminate potential carryover effect from the previous stimulation.

This study aims to investigate the neuropsychological effect of low frequency stimulation of the nucleus basalis of Meynert (NBM) in advanced Parkinson's disease (PD) patients, who were previously treated with deep brain stimulation (DBS) of the globus pallidus interna (GPi).

ELIGIBILITY:
Inclusion Criteria:

* Patients with GPi stimulation, with the NBM within the vicinity of the electric field of at least one DBS electrode.
* Patients should be able to give informed consent
* Patients should be on a stable medication regimen for at least 4 weeks

Exclusion Criteria:

* any unstable internal disease
* Subject with significant worsening of motor function during the pilot screening study, which is indicated by an increase of the UPDRS part III score more than 30%, will not continue to the crossover trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in global cognitive function measured by the Scales for Outcomes in Parkinson's disease-Cognition (SCOPA-COG) | 2 weeks of the crossover trial phase

SECONDARY OUTCOMES:
Changes of Unified Parkinson's Disease Rating Scale (UPDRS) part 3 | 3 days of the screening phase
Changes of the power of background EEG frequencies | 2 weeks of the crossover trial phase
Score changes of stroop test | 2 weeks of the crossover trial phase
Score changes of the Trail Making test | 2 weeks of the crossover trial phase
Score changes of the digit span test of Wechsler Adult Intelligence Scale III | 2 weeks of the crossover trial phase
Score changes of the symbol digit modality test (SDMT) | 2 weeks of the crossover trial phase
Score changes of the Hospital Anxiety and Depression Scale | 2 weeks of the crossover trial phase
Score changes of the Apathy Evaluation Scale | 2 weeks of the crossover trial phase

CONTACTS AND LOCATIONS:
Overall Officials: Teus van Laar, Prof. Dr., Principal Investigator — Department of Neurology, University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided